CLINICAL TRIAL: NCT05447390
Title: Evaluation of the Strength of Handgrip in Patients With Pulmonary Artery Hypertension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Serdar Kula, M.D, Professor, Gazi University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022-397
Record Dates: First submitted 2022-06-28; First posted 2022-07-07 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Pulmonary Hypertension
Keywords: handgrip; functional status
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Intervention Model Description: This study includes 15 patients diagnosed with Pulmonary Hypertension in Gazi Medical School Hospital Department of Pediatric Cardiology and 40 healthy children who applied to Gazi University Medical School Pediatric Cardiology Clinic
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pulmonary Hypertension (Active Comparator)
  Interventions: Diagnostic Test: Handgrip strength test
- Healthy Control (Active Comparator)
  Interventions: Diagnostic Test: Handgrip strength test

INTERVENTIONS:
Diagnostic Test: Handgrip strength test — The Jamar Hydraulic Hand Dynamometer device is used for measuring the handgrip strength test

SUMMARY:
Our study aims to investigate the changes in muscle strength and muscle mass in PAH patients compared to healthy individuals and determine its effects on prognosis.

Further categorization of PAH patients based on their NYHA class will help determine if their handgrip strength decreases while progressing from NYHA class 1 to 4. This in turn allows us to examine if the handgrip test can be considered as an alternative to a 6-minute walking test (6MWT).

The Jamar Hydraulic Hand Dynamometer device in our hospital is used for measuring the handgrip strength test.

The data of the included subjects in this study are obtained and recorded from the existing files. Also, the handgrip strength test data will be recorded after the investigation

DETAILED DESCRIPTION:
In our study, dynamometer tests will be applied to approximately 15 patients diagnosed with PAH. For control purposes, a hand dynamometer test will be applied to 40 healthy children. Patients' age, gender, weight, height, NYHA class, used medications, complete blood count (Hb, Hct, MCV, RDW), BNP, Troponin-t, biochemical parameters, catheterization findings at diagnosis, Echocardiographic findings (Tricuspid Annular Plane Systolic Excursion-TAPSE), Right Ventricular End Systolic Remodeling Index (RVES-RI), Pulmonary Artery acceleration Time (PAaccT), Tricuspid Velocity Time Integral (TR-VTI), RV area, RV length, Right Ventricular Load Adaptation Index (RV LAI), congenital heart disease and whether there is a shunt recorded or not. Patients are informed about the test before the dynamometer test. This may affect the integrity and accuracy of test results. To prevent such inaccuracies, the test will be performed on patients' both hands and the results are not recorded. Patients are asked to sit in a specific position. That is to sit upright with their elbows flexed 90° and the palms facing inwards (medially). Then, the test is performed 3 times with both hands. The results are recorded as the average of all the trials for dominant and non-dominant hands separately. The length of patients' hands is also measured. With the help of this test,it is possible to measure the difference in handgrip strength between healthy subjects and PAH patients. Additionally, patients are divided into 4 groups based on their NYHA classes. This will investigate if the patients' handgrip strength decreases as progress from NYHA class 1 to 4

ELIGIBILITY:
Inclusion Criteria:

Pulmonary Hypertension Group:

* Diagnosed with Pulmonary Hypertension and attending the clinic for follow-ups.
* Older than 5 years.

Healthy Control Group

* Individuals without any known diseases, structural Cardiac anomalies, familial history of heart diseases and sudden death.
* Older than 5 years.

Exclusion Criteria:

Volunteers' Rejection Criteria:

* Younger than 5 years.
* Mental state disorders which will cause inaccuracies in the study's

  i. Volunteers' Dismissal Criteria:
* Inadaptation to the study's steps.
* If subjects become reluctant to continue with the study.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 55 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the strength of handgrip in patients with pulmonary artery hypertension | Baseline
  Investigate and evaluate of the strength of handgrip in patients with pulmonary artery hypertension with hand dynamometer compared to healthy individuals.

SECONDARY OUTCOMES:
Evaluation of the strength of handgrip in patients with pulmonary artery hypertension | Baseline
  Further categorization of PAH patients based on their NYHA class will help determine if their handgrip strength decreases while progressing from NYHA class 1 to 4. This in turn allows us to examine if the handgrip test can be considered as an alternative to a 6-minute walking test (6MWT).

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University School of Medicine, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hansmann G, Koestenberger M, Alastalo TP, Apitz C, Austin ED, Bonnet D, Budts W, D'Alto M, Gatzoulis MA, Hasan BS, Kozlik-Feldmann R, Kumar RK, Lammers AE, Latus H, Michel-Behnke I, Miera O, Morrell NW, Pieles G, Quandt D, Sallmon H, Schranz D, Tran-Lundmark K, Tulloh RMR, Warnecke G, Wahlander H, Weber SC, Zartner P. 2019 updated consensus statement on the diagnosis and treatment of pediatric pulmonary hypertension: The European Pediatric Pulmonary Vascular Disease Network (EPPVDN), endorsed by AEPC, ESPR and ISHLT. J Heart Lung Transplant. 2019 Sep;38(9):879-901. doi: 10.1016/j.healun.2019.06.022. Epub 2019 Jun 21. PMID 31495407
- [Background] Kula S, Pektas A. A review of pediatric pulmonary hypertension with new guidelines. Turk J Med Sci. 2017 Apr 18;47(2):375-380. doi: 10.3906/sag-1605-172. PMID 28425226
- [Background] Di Rienzo A, Felicetti L, Novelletto A, Forteleoni G, Colombo B. Frequency and types of deletional alpha+-thalassemia in northern Sardinia. Hum Genet. 1985;71(2):147-9. doi: 10.1007/BF00283371. PMID 2995236
- [Background] Neidenbach RC, Oberhoffer R, Pieper L, Freilinger S, Ewert P, Kaemmerer H, Nagdyman N, Hager A, Muller J. The value of hand grip strength (HGS) as a diagnostic and prognostic biomarker in congenital heart disease. Cardiovasc Diagn Ther. 2019 Oct;9(Suppl 2):S187-S197. doi: 10.21037/cdt.2019.09.16. PMID 31737527
- [Background] Mathiowetz V, Wiemer DM, Federman SM. Grip and pinch strength: norms for 6- to 19-year-olds. Am J Occup Ther. 1986 Oct;40(10):705-11. doi: 10.5014/ajot.40.10.705. PMID 3777107
- [Background] Hager-Ross C, Rosblad B. Norms for grip strength in children aged 4-16 years. Acta Paediatr. 2002;91(6):617-25. doi: 10.1080/080352502760068990. PMID 12162590
- [Background] Ploegmakers JJ, Hepping AM, Geertzen JH, Bulstra SK, Stevens M. Grip strength is strongly associated with height, weight and gender in childhood: a cross sectional study of 2241 children and adolescents providing reference values. J Physiother. 2013 Dec;59(4):255-61. doi: 10.1016/S1836-9553(13)70202-9. PMID 24287219